CLINICAL TRIAL: NCT05238922
Title: A Phase 1, Open-Label, Multicenter Study of INCB123667 as Monotherapy and in Combination With Anticancer Therapies in Participants With Selected Advanced Solid Tumors
Brief Title: Study of INCB123667 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB 123667-101; 2021-005357-91 (EudraCT Number)
Record Dates: First submitted 2022-01-31; First posted 2022-02-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors
Keywords: advanced solid tumors; metastatic solid tumors; Gynecological Tumors,; GI Tumors,; Breast Cancer,; Tumor Agnostic; cyclin E1 gene; epithelial ovarian carcinoma; fallopian carcinoma; primary peritoneal carcinoma; clear cell ovarian cancer; endometrial adenocarcinoma; uterine carcinosarcoma; uterine papillary serous carcinoma; gastrointestinal tumors; gastric adenocarcinomas; GEJ adenocarcinomas; esophageal adenocarcinomas
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ovarian Epithelial; Digestive System Neoplasms | interventions — palbociclib; Bevacizumab; olaparib; Paclitaxel; ribociclib; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Part 1a and 2a will be dose escalation using a statistical hybrid design to identify the RDE(s). Parts 1b and 2b will consist of dose expansion to better characterize the safety, tolerability, PK, pharmacodynamics, and preliminary antitumor activity of INCB123667 as monotherapy or in combination with anticancer therapies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (21):
- Phase 1a Dose Escalation (Experimental): INCB123667 will be administered at a protocol defined starting regimen once daily (QD) orally in 28-day cycles.
  Subsequent dose regimens will be determined during study conduct.
  Interventions: Drug: INCB0123667
- Phase 1b: Dose Expansion Cohort Disease Group 1 (Experimental): INCB123667 will be administered at the recommended dose or doses for expansion (RDE[s]) for advanced or metastatic solid tumors. Participants with gynecologic tumors (epithelial ovarian/fallopian/primary peritoneal carcinoma) will enroll in this group.
  Interventions: Drug: INCB0123667
- Phase 1b: Dose Expansion Cohort Disease Group 2 (Experimental): INCB123667 will be administered at the recommended dose or doses for expansion (RDE[s]) for advanced or metastatic solid tumors. Participants with Endometrial/Uterine cancer will enroll in this group.
  Interventions: Drug: INCB0123667
- Phase 1b: Dose Expansion Cohort Disease Group 3 (Experimental): INCB123667 will be administered at the recommended dose or doses for expansion (RDE[s]) for advanced or metastatic solid tumors. Participants with gastric, Gastro Esophageal Junction (GEJ), and esophageal adenocarcinomas will enroll in this group.
  Interventions: Drug: INCB0123667
- Phase 1b: Dose Expansion Cohort Disease Group 4 (Experimental): INCB123667 will be administered at the recommended dose or doses for expansion (RDE[s]) for advanced or metastatic solid tumors. Participants with Triple Negative Breast Cancer(TNBC) will enroll in this group.
  Interventions: Drug: INCB0123667
- Phase 1b: Dose Expansion Cohort Disease Group 5 (Experimental): INCB123667 will be administered at the recommended dose or doses for expansion (RDE[s]) for advanced or metastatic solid tumors. Participants with HR+/HER2- breast cancer who have had disease progression on or been intolerant of a CDK4/6 inhibitor will enroll in this group.
  Interventions: Drug: INCB0123667
- Phase 1b: Dose Expansion Cohort Disease Group 6 (Experimental): INCB123667 will be administered at the recommended dose or doses for expansion (RDE[s]) for advanced or metastatic solid tumors will enroll in this group.
  Interventions: Drug: INCB0123667
- Phase 2a Dose Escalation Treatment Group A (TGA) (Experimental): INCB123667 administered in combination with palbociclib at the recommended doses in participants with HR+/HER2- breast cancer and in participants with a different tumor as defined in the protocol.
  Interventions: Drug: INCB0123667; Drug: Palbociclib
- Phase 2a Dose Escalation Treatment Group B (TGB) (Experimental): INCB123667 administered in combination with palbociclib and fulvestrant at the recommended doses in participants with HR+/HER2- breast cancer as defined in the protocol.
  Interventions: Drug: INCB0123667; Drug: Palbociclib; Drug: Fulvestrant
- Phase 2a Dose Escalation Treatment Group C (TGC) (Experimental): INCB123667 administered in combination with ribociclib at the recommended doses in participants with HR+/HER2- breast cancer and in participants with a different tumor as defined in the protocol.
  Interventions: Drug: INCB0123667; Drug: Ribociclib
- Phase 2a Dose Escalation Treatment Group D (TGD) (Experimental): INCB123667 administered in combination with ribociclib and fulvestrant at the recommended doses in participants with HR+/HER2- breast cancer as defined in the protocol.
  Interventions: Drug: INCB0123667; Drug: Ribociclib; Drug: Fulvestrant
- Phase 2a Dose Escalation Treatment Group E (TGE) (Experimental): INCB123667 administered in combination with bevacizumab at the recommended doses in participants with HR+/HER2- breast cancer and in participants with a different tumor as defined in the protocol.
  Interventions: Drug: INCB0123667; Drug: Bevacizumab
- Phase 2a Dose Escalation Treatment Group F (TGF) (Experimental): INCB123667 administered in combination with olaparib at the recommended doses in participants with HR+/HER2- breast cancer and in participants with a different tumor as defined in the protocol.
  Interventions: Drug: INCB0123667; Drug: Olaparib
- Phase 2a Dose Escalation Treatment Group G (TGG) (Experimental): INCB123667 administered in combination with paclitaxel at the recommended doses in participants with HR+/HER2- breast cancer and in participants with a different tumor as defined in the protocol.
  Interventions: Drug: INCB0123667; Drug: Paclitaxel
- Phase 2b Dose Expansion Treatment Group H (TGH) (Experimental): INCB123667 administered in combination with palbociclib at the recommended doses in participants with HR+/HER2- breast cancer and in participants with a different tumor as defined in the protocol.
  Interventions: Drug: INCB0123667; Drug: Palbociclib
- Phase 2b Dose Expansion Treatment Group I (TGI) (Experimental): INCB123667 administered in combination with palbociclib and fulvestrant at the recommended doses in participants with HR+/HER2- breast cancer as defined in the protocol
  Interventions: Drug: INCB0123667; Drug: Palbociclib; Drug: Fulvestrant
- Phase 2b Dose Expansion Treatment Group J (TGJ) (Experimental): INCB123667 administered in combination with ribociclib at the recommended doses in participants with HR+/HER2- breast cancer and in participants with a different tumor as defined in the protocol.
  Interventions: Drug: INCB0123667; Drug: Ribociclib
- Phase 2b Dose Expansion Treatment Group K (TGK) (Experimental): INCB123667 administered in combination with ribociclib and fulvestrant at the recommended doses in participants with HR+/HER2- breast cancer as defined in the protocol.
  Interventions: Drug: INCB0123667; Drug: Ribociclib; Drug: Fulvestrant
- Phase 2b Dose Expansion Treatment Group L (TGL) (Experimental): INCB123667 administered in combination with bevacizumab at the recommended doses in participants with gynecologic tumors (epithelial ovarian/fallopian/primary peritoneal carcinoma) as defined by the protocol.
  Interventions: Drug: INCB0123667; Drug: Bevacizumab
- Phase 2b Dose Expansion Treatment Group M (TGM) (Experimental): INCB123667 administered in combination with olaparib at the recommended doses in participants with gynecologic tumors (epithelial ovarian/fallopian/primary peritoneal carcinoma) as defined by the protocol.
  Interventions: Drug: INCB0123667; Drug: Olaparib
- Phase 2b Dose Expansion Treatment Group N (TGN) (Experimental): INCB123667 administered in combination with weekly paclitaxel at the recommended doses in participants with gynecologic tumors (epithelial ovarian/fallopian/primary peritoneal carcinoma) as defined by the protocol.
  Interventions: Drug: INCB0123667; Drug: Paclitaxel

INTERVENTIONS:
Drug: INCB0123667 — 25 mg tablets
Drug: Palbociclib — Palbociclib will be administered at protocol defined dose.
  Arms: Phase 2a Dose Escalation Treatment Group A (TGA); Phase 2a Dose Escalation Treatment Group B (TGB); Phase 2b Dose Expansion Treatment Group H (TGH); Phase 2b Dose Expansion Treatment Group I (TGI)
Drug: Bevacizumab — Bevacizumab will be administered at protocol defined dose.
  Arms: Phase 2a Dose Escalation Treatment Group E (TGE); Phase 2b Dose Expansion Treatment Group L (TGL)
Drug: Olaparib — Olaparib will be administered at protocol defined dose.
  Arms: Phase 2a Dose Escalation Treatment Group F (TGF); Phase 2b Dose Expansion Treatment Group M (TGM)
Drug: Paclitaxel — Paclitaxel will be administered at protocol defined dose.
  Arms: Phase 2a Dose Escalation Treatment Group G (TGG); Phase 2b Dose Expansion Treatment Group N (TGN)
Drug: Ribociclib — Ribociclib will be administered at protocol defined dose.
  Arms: Phase 2a Dose Escalation Treatment Group C (TGC); Phase 2a Dose Escalation Treatment Group D (TGD); Phase 2b Dose Expansion Treatment Group J (TGJ); Phase 2b Dose Expansion Treatment Group K (TGK)
Drug: Fulvestrant — Fulvestrant will be administered at protocol defined dose.
  Arms: Phase 2a Dose Escalation Treatment Group B (TGB); Phase 2a Dose Escalation Treatment Group D (TGD); Phase 2b Dose Expansion Treatment Group I (TGI); Phase 2b Dose Expansion Treatment Group K (TGK)

SUMMARY:
This is an open-label, dose-escalation and dose-expansion study to determine the safety, tolerability, PK, pharmacodynamics, and preliminary efficacy of INCB123667 when administered as monotherapy and in combination with anticancer therapies in participants with selected advanced or metastatic solid tumors. This study will consist of 2 parts. In Part 1, INCB123667 will be administered as monotherapy and in Part 2, INCB123667 will be administered in combination with anticancer therapies of interest. Each part will comprise a dose escalation portion (Parts 1a and 2a, respectively) and a dose-expansion portion (Parts 1b and 2b, respectively).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older at the time of the signing of the ICF.
* Life expectancy greater than 12 weeks.
* ECOG performance status score of 0 or 1.
* Disease progression on prior standard treatment, intolerance to or ineligibility for standard treatment, or no available treatment to improve the disease outcome.
* Availability of a baseline archival tumor specimen or willingness to undergo a pretreatment and an on-treatment tumor biopsy.

For Part 1:

Participants in Part 1A (dose escalation): Histologically or cytologically confirmed advanced or metastatic solid tumors.

Participants in Part 1B (dose expansion):

* Disease Group 1: Ovarian/Fallopian/Primary Peritoneal Cancer
* Disease Group 2: Endometrial/Uterine Cancer
* Disease Group 3: Gastric, GEJ, and esophageal carcinomas
* Disease Group 4: TNBC
* Disease Group 5: HR+/HER2- breast cancer
* Disease Group 6: Other tumor indications excluding bone cancers

For Part 2:

Participants in Part 2A (dose escalation): Histologically or cytologically confirmed advanced or metastatic solid tumors.

* TGA, TGC, TGE, TGF, and TGG: Participants with HR+/HER2- breast cancer or participants with a different tumor.
* TGB and TGD: Participants with HR+/HER2- breast cancer.

Participants in Part 2b (dose expansion):

* TGH and TGJ:

  * Participants with HR+/HER2- breast cancer.
  * Participants with any other advanced or metastatic solid tumor.
* TGI and TGK:

  • Participants with HR+/HER2- breast cancer.
* TGL, TGM and TGN:

  • Participants with advanced or metastatic epithelial ovarian/fallopian/primary peritoneal carcinoma.
* Measurable lesions by CT or MRI based on RECIST v1.1 criteria.

Exclusion Criteria:

* History of clinically significant or uncontrolled cardiac disease.
* History or presence of an ECG abnormality that, in the investigator's opinion, is clinically meaningful.
* Presence of chronic or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment.
* Untreated brain or central nervous system (CNS) metastases or brain or CNS metastases that have progressed.
* Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of the first dose of study drug.
* Specific laboratory values.
* Significant concurrent, uncontrolled medical conditions, including but not limited to Hepatic and Gastrointestinal.
* Has not recovered to ≤ Grade 1 from toxic effects of prior therapy and/or complications from prior surgical intervention before starting study drug.
* Prior treatment with any CDK2 inhibitor.
* Any change in endocrine therapy within 5 half-lives or 28 days (whichever is shorter) before the first dose of study drug or any administration of targeted therapy, antibody, or hypomethylating agent to treat the participant's disease within 5 half-lives or 28 days (whichever is shorter) before the first dose of study drug.
* Any major surgery within 28 days before the first dose of study drug.
* Any prior radiation therapy within 28 days before the first dose of study drug.
* Undergoing treatment with another investigational medication or having been treated with an investigational medication within 5 half-lives or 28 days (whichever is shorter) before the first dose of study drug.
* Active HBV or HCV infection that requires treatment.
* Known history of HIV.
* Known hypersensitivity or severe reaction to any component of study treatment or formulation components.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 604 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2027-07-27 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Part 1A : Occurrence of Dose Limiting Toxicities (DLTs) | Up to Day 28
  Toxicities occurring during the first treatment cycle, Part 1a, will define tolerability. DLTs will be assessed for severity by the investigator using CTCAE v5.0 criteria.
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to 12 months
  TEAE is any Adverse Event (AE) either reported for the first time or worsening of a pre-existing event after first dose of study drug.
Number of Participants with Dose Interruptions due to TEAE | Up to 12 months
  Participants will receive dose reductions of INCB123667 according to lab guidelines. Treatment may be delayed for up to 2 weeks to allow for resolution of toxicity.
Number of Participants who Undergo Dose Reductions due to TEAE | Up to 12 months
  Participants will receive dose reductions according to lab guidelines. Treatment may be delayed for up to 2 weeks to allow for resolution of toxicity.
Number of Participants Discontinue study due to TEAE | Up to 12 months
  TEAE is defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
PK parameters: Cmax | Cycle 1 Days 1, 2, 8 and 9; Cycle 2 Day 1; Cycles 3 through 9 Day 1 (each cycle is 28 days)
  Defines as the maximum (peak) plasma drug concentration
PK parameters: tmax | Cycle 1 Days 1, 2, 8 and 9; Cycle 2 Day 1; Cycles 3 through 9 Day 1 (each cycle is 28 days)
  Defined as the time to reach maximum (peak) plasma concentration following drug administration
PK parameters: Ctau | Cycle 1 Days 1, 2, 8 and 9; Cycle 2 Day 1; Cycles 3 through 9 Day 1 (each cycle is 28 days)
  Ctau is defined as concentration at the end of the dosing interval
PK Parameters: AUC | Cycle 1 Days 1, 2, 8 and 9; Cycle 2 Day 1; Cycles 3 through 9 Day 1 (each cycle is 28 days)
  Defined as the area under the plasma concentration-time curve
PK Parameters: CL/F | Cycle 1 Days 1, 2, 8 and 9; Cycle 2 Day 1; Cycles 3 through 9 Day 1 (each cycle is 28 days)
  Defined as the apparent total body clearance of the drug from plasma
PK Parameters: Vz/F | Cycle 1 Days 1, 2, 8 and 9; Cycle 2 Day 1; Cycles 3 through 9 Day 1 (each cycle is 28 days)
  Defined as apparent volume of distribution during terminal phase
PK Parameters: t1/2 | Cycle 1 Days 1, 2, 8 and 9; Cycle 2 Day 1; Cycles 3 through 9 Day 1 (each cycle is 28 days)
  Defined as Elimination half-life (to be used in one-or noncompartmental model)
Objective Response Rate (ORR) | Up to 12 months
  Defined as having a best overall Complete Response (CR) or Partial Response (PR), as determined by the investigator by radiographic disease assessment according to RECIST v1.1.
Disease Control | Up to 12 months
  Defined as having a best overall response of CR, PR, or Stable Disease (SD) as determined by the investigator by radiographic disease assessment according to RECIST v1.1.
Duration of Response (DOR) | Up to 12 months
  Defined as the time from earliest date of disease response (Completed Response or Partial Response) until earliest date of disease progression as determined by the investigator by radiographic disease assessment according to RECIST v1.1 or death due to any cause if occurring sooner than progression.

CONTACTS AND LOCATIONS:
Overall Officials: Liz Croft, MD, Study Director — Incyte Corporation
Locations (46):
- United States (21):
  - City of Hope Medical Center, Duarte, California
  - City of Hope-Lennar Foundation Cancer Center, Irvine, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Mount Sinai Medical Center Comprehensive Cancer Center, Miami Beach, Florida
  - Emory University, Atlanta, Georgia
  - University of Kansas Cancer Center, Westwood, Kansas
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian/Weill Cornell, New York, New York
  - Ny Cancer and Blood Specialists, Shirley, New York
  - Carolina Bio-Oncology Institute, Pllc, Huntersville, North Carolina
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute Cancer Services, Pittsburgh, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology, Austin, Texas
  - Texas Oncology-Fort Worth South Henderson, Fort Worth, Texas
  - Virginia Cancer Institute, Fairfax, Virginia
  - University of Wisconsin, Madison, Wisconsin
- France (5):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
  - Universitaire Du Cancer de Toulouse Institut Claudius Regaud Iuct-Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Italy (5):
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Istituto Nazionale Tumori Irccs Fondazione Pascale, Naples
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Rome
  - Irccs Istituto Clinico Humanitas, Rozzano
  - Centro Ricerche Cliniche Di Verona, Verona
- Japan (5):
  - Aichi Cancer Center Hospital, Aichi
  - National Cancer Center Hospital East, Chiba-ken
  - Saitama Medical University International Medical Center, Hidaka-shi
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of Jfcr, Tokyo
- Netherlands (2):
  - Netherlands Cancer Institute Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam
  - Erasmus Medical Center, Rotterdam
- Panoncology Trials Pan American Center For Oncology Trials, Llc, Rio Piedras, Puerto Rico
- Switzerland (3):
  - Oncological Institute of Southern Switzerland, Bellinzona
  - Inselspital Universitatsklinik Fur Medizinische Onkologie, Bern
  - Centre Hospitalier Universitaire Vaudois (Chuv), Lausanne
- United Kingdom (4):
  - Guys Hospital, London
  - Imperial College Healthcare Nhs Trust - Hammersmith Hospital, London
  - The Christie Nhs Foundation Trust Uk, Manchester
  - Northern Centre For Cancer Care, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study of INCB123667 in Subjects with Advanced Solid Tumors — https://incyteclinicaltrials.com/studies/incb-123667-101